CLINICAL TRIAL: NCT01712737
Title: The Effects of Ad Libitum Pre-Meal Raisin Snack on Satiety and Food Intake in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Mount Saint Vincent University (Other); Toronto Metropolitan University (Other); California Raisin Marketing Board (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Raisins_part1_UofT
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Food Intake Regulation
Keywords: raisins, grapes, snacks, appetite, food intake
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Snack foods: raisins (Experimental): children were given ad libitum access to raisins for 15 min
  Interventions: Other: Dietary intervention
- Snack foods: grapes (Experimental): children were given ad libitum access to grapes for 15 min
  Interventions: Other: Dietary intervention
- Snack foods: a mix of almonds with raisins (Experimental): children were given ad libitum access to a mix of almonds with raisins for 15 min
  Interventions: Other: Dietary intervention
- Water control (Experimental): children were given ad libitum access to water
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention

SUMMARY:
No studies have reported the effect of pre-meal snacking on raisins compared to other commonly consumed snacks on energy intake in children. Therefore, the objective of the current study was to examine appetite and energy intake following consumption of ad libitum snack of raisins, grapes or mix of almonds and raisins, compared with a water control, on appetite and food intake 30 min later in 8 - 11 y old normal weight children. The investigators hypothesized that raisins would lower subsequent energy intake in children and reduce hunger.

ELIGIBILITY:
Inclusion Criteria: healthy boys and girls between 8-11 y Exclusion criteria: learning and behavioral problems

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
ad libitum snack intake (kcal) | 15 min
ad libitum pizza intake (kcal) | at 30 min after treatment

SECONDARY OUTCOMES:
subjective appetite | 0-105 min

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Anderson, PhD, Principal Investigator — University of Toronto